CLINICAL TRIAL: NCT06631170
Title: A Phase 3 Multicenter, Double-blind, Vehicle-controlled Brigding Study to Evaluate the Efficacy and Safety of Roflumilast Cream 0.15% (ZORYVE®) in the Treatment of Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Efficacy and Safety of Roflumilast Cream in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HDM3014-2-301
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Roflumilast cream; Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Roflumilast cream 0.15% (Experimental): Active comparator
  Interventions: Drug: Roflumilast Cream 0.15%
- Vehicle cream (Placebo Comparator): Placebo comparator
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Roflumilast Cream 0.15% — Roflumilast cream 0.15% is applied once daily for 4 weeks
  Arms: Roflumilast cream 0.15%
Drug: Vehicle cream — Vehicle cream is applied once daily for 4 weeks
  Arms: Vehicle cream

SUMMARY:
This study will assess the safety and efficacy of Roflumilast cream versus vehicle applied once a day for 4 weeks by subjects with atopic dermatitis.

DETAILED DESCRIPTION:
This is a parallel group, double blind, vehicle-controlled study in which Roflumilast cream or vehicle is applied once daily for 4 weeks to subjects with mild or moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 6 years at screening.
2. Diagnosed with atopic dermatitis (AD) for at least 6 months for subjects aged ≥18 years and 3 months for subjects aged 6~17 years at screening.
3. Have stable disease for the past 4 weeks prior to screening.
4. Have mild or moderate AD at baseline.
5. Have BSA affected by AD of 3%-20% at baseline.
6. Women of childbearing potential (WOCBP) have a negative pregnancy blood test at screening and a negative urine pregnancy test at baseline. WOCBP must have taken and agree to continue taking highly effective contraceptive measures from 4 weeks before the first dose to 2 months after the last dose.
7. Being in good health as judged by the Investigator.
8. Subjects voluntarily participate in the study and sign the ICF before the start of study-related activities.

Exclusion Criteria:

1. Subjects with any serious medical condition or clinically significant abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator.
2. Previous treatment with roflumilast cream.
3. Use of systemic treatments that affect the efficacy assessment of AD 4 weeks or 5 half-lives (whichever is longer) prior to the first dose.
4. Use of topical treatments that affect the efficacy assessment of AD 2 weeks prior to the first dose.
5. Use of phototherapy, tanning beds, or any other light-emitting devices within 4 weeks prior to the first dose.
6. Female subjects who are pregnant or breastfeeding, or plan to become pregnant or breastfeed during the study.
7. Subjects with a history of chronic alcohol or drug abuse within 6 months prior to Screening.
8. Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members of enrolled subjects living in the same house.
9. Subjects/legal guardians who are unable to communicate, understand the study, or other situations deemed inappropriate for participation in a clinical trial by the investigator.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-07-13 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with vIGA-AD success | Baseline, week 4
  The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear). IGA sucess is defined as a vIGA-AD score of 'clear' or 'almost clear' plus at least 2-grade improvement from baseline

SECONDARY OUTCOMES:
In subjects with moderate AD severity (vIGA-AD score of 3) at baseline, percentage of subjects with vIGA-AD success | Baseline, week 4
  The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear).
Percentage of subjects with vIGA-AD of "clear" or "almost clear" | Baseline, week 4
  The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear).
In subjects with WI-NRS ≥ 4 at baseline, percentage of subjects with ≥ 4 point reduction in WI-NRS | Baseline, week 4
  The Worst Itch Numerical Rating Scale (WI-NRS) will be determined by the subject's recording of daily assessment of worst itch over the past 24 hours. The scale is from '0 to 10' ("no itch" to "worst itch imaginable" or "worst imaginable itch").
Percentage of subjects with at least 75% reduction in the Eczema Area and Severity Index (EASI-75) | Baseline, week 4
  EASI combines the assessment of the severity of lesions and the area affected into a single total score in the range 0 (no disease) to 72 (maximal disease). Four anatomic sites-head, upper extremities, trunk, and lower extremities-are assessed for erythema, induration/infiltration (papules), excoriation, and lichenification as seen on the day of the examination. To calculate the EASI, the sum of the severity rating (0 to 3 with 3 being the most severe) for four clinical signs are multiplied with the numerical value of the area affected and with the percentage of the four body areas.
Safety: treatment emergence adverse events | Up to 4 weeks
  Incidence, severity, and causal relationship of treatment emergence adverse events (TEAE), TEAEs leading to withdrawal and death.
Trough concentration (Ctrough) | Week 2, week 4
  Trough concentration of plasma roflumilast and its N-oxide

CONTACTS AND LOCATIONS:
Locations (61):
- China (61):
  - The Second affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Aerospace General Hospital, Beijing, Beijing Municipality
  - Beijing Children's Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, CMU, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Chongqing Medical University Affiliated Second Hospital, Chongqing, Chongqing Municipality
  - People's Hospital Affiliated to Chongqing Three Gorges Medical College, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The Second affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - The Sixth People's Hospital of Dongguan, Dongguan, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Union Shenzhen Hospital, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The Fifth People's Hospital of Hainan Province, Haikou, Hainan
  - Kunming Children's Hospital, Kunming, Hainan
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - TCM Hospital of Shi Jia Zhuang City, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The Second Hospital affiliated to Henan University of Science and Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Henan Children's Hospital Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - Hunan Children's Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital, Changsha, Hunan
  - Sir Run Run Hospital Nanjing Medical University, Nanjing, Jiangsu
  - J.Y Hospital of TCM, Wuxi, Jiangsu
  - People's hospital of Wuxi, Wuxi, Jiangsu
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - The Second affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Dalian Dermatology Hospital, Dalian, Liaoning
  - Dalian Municipal Women and Children's Medical Center, Dalian, Liaoning
  - Panjin Liaohe Oilfield Gem Flower Hospital, Panjin, Liaoning
  - The First affiliated Hospital of Baotou College, Baotou, Neimenggu
  - Jinan Central Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Hiser Medical Center of Qingdao, Qingdao, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Children's Hospital, Shanghai, Shanghai Municipality
  - The Second affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The Second Hospital of Jiaxing, Jiaxing, Zhejiang
  - The Second Hospital of Ningbo, Ningbo, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No